CLINICAL TRIAL: NCT05246046
Title: Pharmacokinetic Study to Compare Tiotropium Easyhaler® Product Variants and Spiriva® 18 µg Capsules Administered Via HandiHaler® in Healthy Volunteers.
Brief Title: Comparison of Tiotropium Absorption From Tiotropium Easyhaler and Spiriva HandiHaler
Acronym: TEMPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3122006
Record Dates: First submitted 2022-02-07; First posted 2022-02-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Hardness

STUDY DESIGN:
Masking Description: Bioanalytical laboratory will be blinded with regard to the sequence of the product administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tiotropium Easyhaler 10 microg/dose, Product variant J (Experimental): Each subject will receive a single dose of 2 inhaled doses from Tiotropium Easyhaler Product variant J in one of the three periods (cross-over). The total dose is 20 micrograms of tiotropium (delivered dose) as Tiotropium Bromide Monohydrate.
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler 10 microg/dose, Product variant K (Experimental): Each subject will receive a single dose of 2 inhaled doses from Tiotropium Easyhaler Product variant K in one of the three periods (cross-over). The total dose is 20 micrograms of tiotropium (delivered dose) as Tiotropium Bromide Monohydrate.
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Spiriva HandiHaler 18 microg/capsule (Active Comparator): Each subject will receive a single dose of 2 inhaled Spiriva capsules via HandiHaler device in one of the three periods (cross-over). The total dose is 20 micrograms of tiotropium (delivered dose) as Tiotropium Bromide Monohydrate.
  Interventions: Drug: Tiotropium Bromide Monohydrate

INTERVENTIONS:
Drug: Tiotropium Bromide Monohydrate — In each period, subjects receive single dose of tiotropium consisting of 2 inhaled doses via Easyhaler or 2 Spiriva capsules inhaled via HandiHaler
  Other Names: Tiotropium Easyhaler 10 microg/dose, inhalation powder, Product variant J; Tiotropium Easyhaler 10 microg/dose, inhalation powder, Product variant K; SPIRIVA® 18 microgram, inhalation powder, hard capsule inhaled via HandiHaler

SUMMARY:
This is a pivotal study to investigate absorption of inhaled tiotropium from 2 Tiotropium Easyhaler product variants and Spiriva capsules inhaled via HandiHaler.

ELIGIBILITY:
Main inclusion criteria:

1. Healthy male and female
2. 18-60 years of age
3. Body mass index 19-30 kg/m2
4. Weight at least 50 kg
5. FEV1 at least 80% of the predicted value measured at screening
6. Written informed consent obtained

Main exclusion criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic, endocrine, neurological or psychiatric disease.
2. Any condition requiring regular concomitant treatment.
3. Any clinically significant abnormal laboratory value or physical finding that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject.
4. Known hypersensitivity to tiotropium bromide, atropine or its derivatives or lactose.
5. Pregnant or lactating females and females of childbearing potential not using contraception of acceptable effectiveness.
6. Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Peak tiotropium concentration in plasma (Cmax) | between 0-72 hours after dosing
Area under the concentration-time curve from time zero to 30 minutes (AUC30 minutes) | between 0-30 minutes after dosing
Area under the concentration-time curve from time zero to 72 hours (AUC72 hours) | between 0-72 hours after dosing

SECONDARY OUTCOMES:
Time to reach peak concentration in plasma (tmax) | between 0-72 hours after dosing

OTHER OUTCOMES:
Adverse events | throughout the study, an average 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orion Corporation Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Clinical Pharmacology Unit, Orion Corporation, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No